CLINICAL TRIAL: NCT01434784
Title: Update of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) Phases I - III
Brief Title: Update of the EORTC QLQ-LC13 Quality of Life Questionnaire
Status: Completed | Type: Observational
Sponsor: Michael Koller (Other)
Collaborators: Hospital of Navarra (Other); Oslo University Hospital (Other); Medical University of Graz (Other); University of Roma La Sapienza (Other); National Taiwan University Hospital (Other); University of Sydney (Other); University of Wuerzburg (Other)
Responsible Party: Sponsor-Investigator, Michael Koller, Prof. Dr., Head of Center for Clinical Studies, University Hospital Regensburg
Organization: University Hospital Regensburg (Other)
Other Study IDs: Koller Lung 03/2010
Record Dates: First submitted 2011-09-12; First posted 2011-09-15 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: lung cancer; quality of life
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Surgery alone: Patients undergoing any kind surgery for lung cancer, no additional surgery, quality of life assessment with the provisional updated lung cancer module within 3 months after surgery
- Surgery in combination with any other tx: Patients undergoing any kind surgery for lung cancer, additional therapy is permitted, quality of life assessment with the provisional updated lung cancer module within 3 months after surgery
- Surgery (late effects): Patients undergoing any kind surgery for lung cancer, additional therapy is permitted, quality of life assessment with the provisional updated lung cancer moduleat least 3 months after surgery and 3 months after any other active treatment
- Chemotherapy alone: Patient undergoing any kind of chemotherapy for lung cancer, no additional therapy, quality of life assessment with the provisional updated lung cancer module during or up to 4 weeks after completion of therapy
- Radiotherapy alone: Patient undergoing radiotherapy for lung cancer, no additional therapy, quality of life assessment with the provisional updated lung cancer module during or up to 3 months after completion of therapy
- Sequential radiochemotherapy: Patient undergoing sequential radiochemotherapy for lung cancer, no surgery, no targeted therapy, quality of life assessment with the provisional updated lung cancer module during or up to 3 months after completion of therapy
- Concurrent radiochemotherapy: Patient undergoing concurrent radiochemotherapy for lung cancer, no surgery, no targeted therapy, quality of life assessment with the provisional updated lung cancer module during or up to 3 months after completion of therapy
- Targeted therapy alone: Patient undergoing targeted therapy for lung cancer, no surgery, no radiochemotherapy , quality of life assessment with the provisional updated lung cancer module during or up to 4 weeks after completion of therapy
- Targeted therapy in combination: Patient undergoing targeted therapy for lung cancer, additional therapies permitted, quality of life assessment with the provisional updated lung cancer module during or up to 3 months after completion of therapy

SUMMARY:
The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) is considered as a standard instrument to assess the quality of life (QL) of lung cancer patients. Since its publication in 1994, major clinical advances have been made. The research objective is to develop a revised lung cancer module that (a) covers all QL aspects relevant in the context of newly available diagnostic and therapeutic options, (b) is applicable in both non-metastatic and metastatic cancers, (c) and covers QL aspects that are generally relevant for patients with lung cancer but are missing in the original module. This project will comprise the first three project phases according to the Module Development Manual (www.eortc.be/qol).

DETAILED DESCRIPTION:
The project follows the EORTC model of module development and covers the first three phases:

Phase I This phase is aimed at compiling an extensive list of quality of life issues relevant for lung cancer patients. The following sources will be used: (1) existing questionnaires on lung cancer and respiratory illnesses, (2) the literature, (3) investigator's brochures (IB) on new drugs, and (4) interviews with health care professionals and patients.

Phase II Phase I data will provide information about the issues that should be included in an improved lung cancer module. These issues are being converted into items that follow the EORTC format with four point response scales ranging from "not at all" to "very much". For the sake of consistency and whenever possible, items of the existing QLC-LC13 will be used or other items will be taken from the Item Bank that currently includes more than 6.000 items. After this stage, the procedure will be formally peer-reviewed by the EORTC QLG Module Development Committee. After approval, the provisional list of items is ready for Phase III.

Phase III The provisional lung cancer module will be pre-tested in an international group of patients with lung cancer. Patients will be first asked to fill in the QLQ-C30 and the provisional revised lung cancer module. After completing the forms, patients will be interviewed with regard to the revised lung cancer module. The interview will identify questionnaire items that patients find annoying, confusing or upsetting. A further issue is relevance: patients should indicate whether there are issues they find irrelevant or whether issues not yet included in the provisional module need to be added. The interviewer, either a physician or a study nurse, will record patients' comments on the debriefing questionnaire.

The sample matrix specifies three main groups according to primary therapy which can be either surgery, radiochemotherapy or targeted therapy.

The singular use or combination of these therapies yields nine subgroups of patients:

1.1 Surgery alone 1.2 Surgery in combination with any other therapy 1.3 Surgery (late effects) 2.1 Chemotherapy alone 2.2 Radiotherapy alone 2.3 Sequential radiochemotherapy 2.4 Concurrent radiochemotherapy 3.1 Targeted therapy alone 3.2 Targeted therapy in combination with any other therapy

The recruitment goal is n = 15 per subgroup, resulting in a total of 135 patients.

Recruitment will take place in the following study regions: English speaking countries including the United Kingdom and Australia; Northern Europe including Norway and Germany; Southern Europe including Italy and Spain; Eastern Europe, and one non-European country (e.g., Taiwan).

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of lung cancer
* informed consent
* capability to respond to a questionnaire and to follow an interview

Exclusion Criteria:

* no informed consent
* lack of capability to respond to a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with confirmed diagnosis of lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Importance of quality of life issues from patients' perspective | in the course or up to three months after having completed therapy
  Importance of quality of life issues are assessed using a four-point scale (1= not at all, 2 = a little, 3 = quite a bit, 4 = very much. Only issues with a mean of > 2 are considered for inclusion in the questionnaire.

SECONDARY OUTCOMES:
Importance of quality of life issues from health care professionals' perspective | in the course or up to three months after patients have completed therapy
  Importance of quality of life issues are assessed using a four-point scale (1= not at all, 2 = a little, 3 = quite a bit, 4 = very much. Only issues with a mean of > 2 are considered for inclusion in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koller, PhD, Principal Investigator — University Hospital Regensburg
Locations (1):
- Center for Clinical Studies, University Hospital Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No